CLINICAL TRIAL: NCT00524719
Title: A Prospective Randomised Trial Comparing Open Reduction and Internal Fixation, Non-Spanning External Fixation, and Closed Reduction With Percutaneous Fixation in Displaced Distal Radius Fractures With Joint Congruity
Brief Title: Comparison of Three Fixation Techniques for Displaced Distal Radius Fractures
Acronym: DRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Principal Investigator, Greg K. Berry, MD, MDCM FRCSC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEN # 05-014
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Distal Radius Fractures
MeSH Terms: conditions — Wrist Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Open, internal fixation volar plate (Active Comparator): Open reduction and internal fixation (ORIF) with volar locked plate
  Interventions: Procedure: Open Reduction and Internal Fixation
- Closed reduction with external fixator (Active Comparator): Surgical procedure - Closed reduction and non-spanning external fixation (Ex-FIX)
  Interventions: Procedure: Non-Spanning External Fixation
- Closed reduction percutaneous pinning (Active Comparator): Surgical procedure - Closed reduction with percutaneous pinning (CRPP) and the application of a cast
  Interventions: Procedure: Closed Reduction with Percutaneous Fixation

INTERVENTIONS:
Procedure: Open Reduction and Internal Fixation — Fixation with volar locked plate
  Arms: Open, internal fixation volar plate
Procedure: Non-Spanning External Fixation — Radio-radial external fixation
  Arms: Closed reduction with external fixator
Procedure: Closed Reduction with Percutaneous Fixation — Percutaneous intrafocal pinning (Kapandji technique)
  Arms: Closed reduction percutaneous pinning

SUMMARY:
Distal radius fractures are the most common fracture to occur in the adult population, and those which are displaced but maintain joint congruity are the most common subtype. Locking-plate technology represents a true advance in the fixation of these fractures, especially in view of the ever increasing incidence of these injuries in an ageing and osteoporotic population throughout Europe and North America. These plates permit rigid fixation, even in osteopenic bone, while avoiding any tethering of soft tissues, as seen with external fixation and percutaneous pinning. For these reasons, this mode of fracture fixation has rapidly gained popularity. Unfortunately, there is presently little evidence to support their use over the more traditional methods of fixation (percutaneous pinning, external fixation). In addition, the technique for their application is more invasive and their cost is considerably greater than these latter two techniques. As such, it is pertinent to evaluate, in a scientifically sound fashion, the outcome of fixation with the three types of implant included in this study. The results of this clinical trial will allow the orthopaedic community to confidently recommend the fixation method which provides the optimal functional, clinical, and radiographic outcome for a patient suffering a displaced distal radius with preserved joint congruity.

Null hypothesis: There is no difference in the functional, clinical, and radiographic outcomes of the three treatment methods.

Hypothesis: Given the locking nature of modern screw-plate constructs, which produce excellent fixation even in osteopenic bone and permit early range of motion exercises; and given that plate fixation, in contrast to external fixation and percutaneous pinning, does not tether muscle, tendon, or capsule; plate fixation with a volar fixed-angle device should permit earlier and more aggressive rehabilitation and more rapid and complete regain of hand and wrist function when compared to stabilization with external fixation or percutaneous pinning.

DETAILED DESCRIPTION:
Fractures of the distal radius, the most common fracture to occur in adults, are increasing in incidence and cost due to ageing of the population and the link with senile osteoporosis. Young adults also suffer these injuries albeit involving higher-energy mechanisms. Closed reduction and casting is often unsuccessful in maintaining adequate alignment and length, both of which are crucial to a successful outcome. Thus, there has been a trend toward surgical treatment of these fractures. In fractures with preserved joint congruity, 3 fixation options exist: percutaneous pinning (Kapandji technique), non-spanning external fixation, and locked-plates. Locked-plates represent a significant advance in the fixation of fractures, especially in osteopenic bone, although their role in distal radius fractures has yet to be defined adequately. The Cochrane Group undertook a meta-analysis of RC trials "to determine when, and if so what type of, surgical intervention is the most appropriate treatment for fractures of the distal radius in adults." The authors concluded: "there is a need for good quality evidence for the surgical management of these fractures." The aim of this randomized clinical trial is to compare the functional, clinical, and radiographic outcomes of these 3 methods. The results will clearly guide surgeons in the choice of optimal technique.

This multicenter prospective randomized trial will involve the Canadian Orthopaedic Trauma Society (COTS), an association of trauma surgeons involved in collaborative outcomes research with a proven track record of research and publication. Patients with a displaced distal radius fracture with joint congruity who meet all eligibility criteria and provide consent to participate will be randomly assigned to reduction and fixation with one of three methods: volar locked-plate, percutaneous pinning and cast (Kapandji intra-focal technique), or non-spanning external fixation. Patients will undergo physiotherapy according to protocols adapted to fixation technique. Evaluation at fixed intervals will include functional, clinical, and radiological parameters. Functional evaluation will include the PRWE, DASH, and SMFA questionnaires. Clinical outcome will evaluate range of motion, pinch and grip strength, and dexterity. Standard radiographic parameters will be measured. The primary outcome measure will be functional outcome as measured with the PRWE. Appropriate statistical analyses will be performed on the data. Sample size calculation reveals the need for 108 patients per treatment arm. A census of the centers committed to the study predicts a 12-18 month recruitment period. Patient follow-up will end at 2 years.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Over 18 years of age with skeletal maturity, and consenting to participate.
2. A displaced distal metaphyseal radius fracture (AO type A2, A3, C1, C2--- appendix 1) with a congruous joint surface (< 2 mm displacement) either before or after closed reduction.
3. 21 days or less between injury and surgery.
4. The patient must be medically fit for anaesthesia.
5. The patient must have the mental faculties to participate in post- operative evaluation.

Patient exclusion criteria:

1. Significant bone disorder (osteomalacia, hyperparathyroidism) which may impair bone healing (not including osteoporosis).
2. Open fracture.
3. Neurovascular injury requiring repair in same limb.
4. Ipsilateral limb injury.
5. Active infection in area of surgical approaches.
6. Prior wrist injury or degenerative condition, or congenital wrist anomaly.

Fracture inclusion criteria:

Patients sustaining a displaced AO type A2 A3 C1 or C2 distal metaphyseal radius fracture with preserved joint congruity before (52) or after closed reduction are eligible for inclusion. Radiographic criteria for an unacceptable closed reduction include:

1. Palmar tilt < 00.
2. Radial inclination < 150.
3. Radial shortening > 5 mm.
4. Articular step or gap > or= 2 mm.

Fracture exclusion criteria:

1. Fractures with apex dorsal angulation ("Smith fracture") will be excluded as they are not amenable to treatment with all three methods.
2. Less than 1 cm of intact volar cortex on the distal fragment as this is the minimum necessary for non-spanning external fixation (40, 48).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2007-01; Primary Completion 2016-12 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Variable: Validated functional outcome tools to be used: patient rated wrist evaluation (PRWE) disability shoulder, arm, hand (DASH) short musculoskeletal functional assessment (SMFA) | 6 weeks; 3,6,12 and 24 months

SECONDARY OUTCOMES:
Secondary Outcome Measures: Clinical outcome: measurement of range of motion (ROM), strength (grip and pinch), and dexterity (Jebsen hand function-checkers sub-test). Radiologic outcome: X-ray parameters | 6 weeks; 3,6,12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Greg K Berry, MD FRCSC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre - Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larsen CF, Lauritsen J. Epidemiology of acute wrist trauma. Int J Epidemiol. 1993 Oct;22(5):911-6. doi: 10.1093/ije/22.5.911. PMID 8282472
- [Background] Nguyen TV, Center JR, Sambrook PN, Eisman JA. Risk factors for proximal humerus, forearm, and wrist fractures in elderly men and women: the Dubbo Osteoporosis Epidemiology Study. Am J Epidemiol. 2001 Mar 15;153(6):587-95. doi: 10.1093/aje/153.6.587. PMID 11257067
- [Background] Cummings SR, Kelsey JL, Nevitt MC, O'Dowd KJ. Epidemiology of osteoporosis and osteoporotic fractures. Epidemiol Rev. 1985;7:178-208. doi: 10.1093/oxfordjournals.epirev.a036281. No abstract available. PMID 3902494
- [Background] Papadimitropoulos EA, Coyte PC, Josse RG, Greenwood CE. Current and projected rates of hip fracture in Canada. CMAJ. 1997 Nov 15;157(10):1357-63. PMID 9371065
- [Background] Goeree R, O'Brien B, Pettit D, Cuddy L, Ferraz M, Adachi JD. An assessment of the burden of illness due to osteoporosis in Canada. J Soc Obstet Gynaecol Can 1996; 18 suppl (July):15-24. 4.
- [Background] Ray NF, Chan JK, Thamer M, Melton LJ 3rd. Medical expenditures for the treatment of osteoporotic fractures in the United States in 1995: report from the National Osteoporosis Foundation. J Bone Miner Res. 1997 Jan;12(1):24-35. doi: 10.1359/jbmr.1997.12.1.24. PMID 9240722
- [Background] van Leeuwen PA, Reynders PA, Rommens PM, Broos PL. Operative treatment of Smith-Goyrand fractures. Injury. 1990 Nov;21(6):358-60. doi: 10.1016/0020-1383(90)90118-e. PMID 2276796
- [Background] Oskam J, Kingma J, Klasen HJ. Fracture of the distal forearm: epidemiological developments in the period 1971-1995. Injury. 1998 Jun;29(5):353-5. doi: 10.1016/s0020-1383(97)00212-x. PMID 9813678
- [Background] Gliatis JD, Plessas SJ, Davis TR. Outcome of distal radial fractures in young adults. J Hand Surg Br. 2000 Dec;25(6):535-43. doi: 10.1054/jhsb.2000.0373. PMID 11106514
- [Background] Szabo RM. Extra-articular fractures of the distal radius. Orthop Clin North Am. 1993 Apr;24(2):229-37. PMID 8479721
- [Background] Kapoor H, Agarwal A, Dhaon BK. Displaced intra-articular fractures of distal radius: a comparative evaluation of results following closed reduction, external fixation and open reduction with internal fixation. Injury. 2000 Mar;31(2):75-9. doi: 10.1016/s0020-1383(99)00207-7. PMID 10748808
- [Background] Kazuki K, Kusunoki M, Yamada J, Yasuda M, Shimazu A. Cineradiographic study of wrist motion after fracture of the distal radius. J Hand Surg Am. 1993 Jan;18(1):41-6. doi: 10.1016/0363-5023(93)90242-U. PMID 8423316
- [Background] McQueen M, Caspers J. Colles fracture: does the anatomical result affect the final function? J Bone Joint Surg Br. 1988 Aug;70(4):649-51. doi: 10.1302/0301-620X.70B4.3403617.
- [Background] Board T, Kocialkowski A, Andrew G. Does Kapandji wiring help in older patients? A retrospective comparative review of displaced intra-articular distal radial fractures in patients over 55 years. Injury. 1999 Dec;30(10):663-9. doi: 10.1016/s0020-1383(99)00167-9. PMID 10707240
- [Background] Stoffelen DV, Broos PL. Closed reduction versus Kapandji-pinning for extra-articular distal radial fractures. J Hand Surg Br. 1999 Feb;24(1):89-91. doi: 10.1016/s0266-7681(99)90045-1. PMID 10190614
- [Background] Jupiter JB, Lipton H. The operative treatment of intraarticular fractures of the distal radius. Clin Orthop Relat Res. 1993 Jul;(292):48-61. PMID 8519137
- [Background] Knirk JL, Jupiter JB. Intra-articular fractures of the distal end of the radius in young adults. J Bone Joint Surg Am. 1986 Jun;68(5):647-59. PMID 3722221
- [Background] Prommersberger KJ, Lanz U. [Biomechanical aspects of malunited distal radius fracture. A review of the literature]. Handchir Mikrochir Plast Chir. 1999 Jul;31(4):221-6. doi: 10.1055/s-1999-13905. German. PMID 10481796
- [Background] Pogue DJ, Viegas SF, Patterson RM, Peterson PD, Jenkins DK, Sweo TD, Hokanson JA. Effects of distal radius fracture malunion on wrist joint mechanics. J Hand Surg Am. 1990 Sep;15(5):721-7. doi: 10.1016/0363-5023(90)90143-f. PMID 2229966
- [Background] Svensson O, Ahrengart L, Ekholm C, Andersson GL, Hoglund M, Jonsson U, Juhlin L, Kopylov P, Lagerstrom C, Lundborg G, Made C, Mallmin H, Raf L, Tornkvist H. [Malpractice in connection with radius fractures must be reduced. Clear guidelines for treatment and follow-up are required]. Lakartidningen. 2000 Apr 12;97(15):1800-4, 1807-9. Swedish. PMID 10815407
- [Background] Fernandez DL. Fractures of the distal radius: operative treatment. Instr Course Lect. 1993;42:73-88. No abstract available. PMID 8463706
- [Background] Hastings H 2nd, Leibovic SJ. Indications and techniques of open reduction. Internal fixation of distal radius fractures. Orthop Clin North Am. 1993 Apr;24(2):309-26. PMID 8479728
- [Background] McMurtry RY, Jupiter JB. Fractures of the distal radius. In: Skeletal Trauma, ed by Browner B, Jupiter J, Levine A, Trafton P. Philadelphia, WB Saunders, 1991, pp 1063-1094
- [Background] Handoll HH, Madhok R. Surgical interventions for treating distal radial fractures in adults. Cochrane Database Syst Rev. 2003;(3):CD003209. doi: 10.1002/14651858.CD003209. PMID 12917953
- [Background] Tornetta P 3rd, Klein DM, Stein AB, McQueen M. Distal radius fracture. J Orthop Trauma. 2002 Sep;16(8):608-11. doi: 10.1097/00005131-200209000-00013. No abstract available. PMID 12352573
- [Background] Kapandji A. [Internal fixation by double intrafocal plate. Functional treatment of non articular fractures of the lower end of the radius (author's transl)]. Ann Chir. 1976 Nov;30(11-12):903-8. No abstract available. French. PMID 1008457
- [Background] Rayhack JM. The history and evolution of percutaneous pinning of displaced distal radius fractures. Orthop Clin North Am. 1993 Apr;24(2):287-300. PMID 8479726
- [Background] Lenoble E, Dumontier C, Goutallier D, Apoil A. Fracture of the distal radius. A prospective comparison between trans-styloid and Kapandji fixations. J Bone Joint Surg Br. 1995 Jul;77(4):562-7. PMID 7615598
- [Background] Peyroux LM, Dunaud JL, Caron M, Ben Slamia I, Kharrat M. The Kapandji technique and its evolution in the treatment of fractures of the distal end of the radius. Report on a series of 159 cases. Ann Chir Main. 1987;6(2):109-22. doi: 10.1016/s0753-9053(87)80023-6. English, French. PMID 3322215
- [Background] Millroy P, Coleman S, Ivers R. The Sauve-Kapandji operation. Technique and results. J Hand Surg Br. 1992 Aug;17(4):411-4. doi: 10.1016/s0266-7681(05)80264-5. PMID 1402268
- [Background] Epinette JA, Lehut JM, Cavenaile M, Bouretz JC, Decoulx J. Pouteau-Colles fracture: double-closed "basket-like" pinning according to Kapandji. Apropos of a homogeneous series of 70 cases. Ann Chir Main. 1982;1(1):71-83. doi: 10.1016/s0753-9053(82)80047-1. English, French. PMID 9303045
- [Background] Greatting MD, Bishop AT. Intrafocal (Kapandji) pinning of unstable fractures of the distal radius. Orthop Clin North Am. 1993 Apr;24(2):301-7. PMID 8479727
- [Background] Dowdy PA, Patterson SD, King GJ, Roth JH, Chess D. Intrafocal (Kapandji) pinning of unstable distal radius fractures: a preliminary report. J Trauma. 1996 Feb;40(2):194-8. doi: 10.1097/00005373-199602000-00004. PMID 8637065
- [Background] Rosenthal AH, Chung KC. Intrafocal pinning of distal radius fractures: a simplified approach. Ann Plast Surg. 2002 Jun;48(6):593-9. doi: 10.1097/00000637-200206000-00005. PMID 12055427
- [Background] Sanders RA, Keppel FL, Waldrop JI. External fixation of distal radial fractures: results and complications. J Hand Surg Am. 1991 May;16(3):385-91. doi: 10.1016/0363-5023(91)90002-s. PMID 1861015
- [Background] Cooney WP. External fixation of distal radial fractures. Clin Orthop Relat Res. 1983 Nov;(180):44-9. PMID 6627796
- [Background] Vaughan PA, Lui SM, Harrington IJ, Maistrelli GL. Treatment of unstable fractures of the distal radius by external fixation. J Bone Joint Surg Br. 1985 May;67(3):385-9. doi: 10.1302/0301-620X.67B3.3997946.
- [Background] Jakim I, Pieterse HS, Sweet MB. External fixation for intra-articular fractures of the distal radius. J Bone Joint Surg Br. 1991 Mar;73(2):302-6. doi: 10.1302/0301-620X.73B2.2005161.
- [Background] McQueen MM, Simpson D, Court-Brown CM. Use of the Hoffman 2 compact external fixator in the treatment of redisplaced unstable distal radial fractures. J Orthop Trauma. 1999 Sep-Oct;13(7):501-5. doi: 10.1097/00005131-199909000-00007. PMID 10513973
- [Background] Kamano M, Honda Y, Kazuki K, Yasuda M. Palmar plating for dorsally displaced fractures of the distal radius. Clin Orthop Relat Res. 2002 Apr;(397):403-8. doi: 10.1097/00003086-200204000-00047. PMID 11953634
- [Background] Jupiter JB. Plate fixation of fractures of the distal aspect of the radius: relative indications. J Orthop Trauma. 1999 Nov;13(8):559-69. doi: 10.1097/00005131-199911000-00009. No abstract available. PMID 10714783
- [Background] Rikli DA, Regazzoni P. Fractures of the distal end of the radius treated by internal fixation and early function. A preliminary report of 20 cases. J Bone Joint Surg Br. 1996 Jul;78(4):588-92. PMID 8682826
- [Background] Hove LM, Nilsen PT, Furnes O, Oulie HE, Solheim E, Molster AO. Open reduction and internal fixation of displaced intraarticular fractures of the distal radius. 31 patients followed for 3-7 years. Acta Orthop Scand. 1997 Feb;68(1):59-63. doi: 10.3109/17453679709003977. PMID 9057570
- [Background] Heim D. [Plate osteosynthesis of distal radius fractures--incidence, indications and results]. Swiss Surg. 2000;6(6):304-14. doi: 10.1024/1023-9332.6.6.304. German. PMID 11142154
- [Background] Campbell DA. Open reduction and internal fixation of intra articular and unstable fractures of the distal radius using the AO distal radius plate. J Hand Surg Br. 2000 Dec;25(6):528-34. doi: 10.1054/jhsb.2000.0485. PMID 11106513
- [Background] Carter PR, Frederick HA, Laseter GF. Open reduction and internal fixation of unstable distal radius fractures with a low-profile plate: a multicenter study of 73 fractures. J Hand Surg Am. 1998 Mar;23(2):300-7. doi: 10.1016/S0363-5023(98)80131-7. PMID 9556273
- [Background] McQueen MM. Redisplaced unstable fractures of the distal radius. A randomised, prospective study of bridging versus non-bridging external fixation. J Bone Joint Surg Br. 1998 Jul;80(4):665-9. doi: 10.1302/0301-620x.80b4.8150. PMID 9699834
- [Background] Franck WM, Dahlen C, Amlang M, Friese F, Zwipp H. [Distal radius fracture--is non-bridging articular external fixator a therapeutic alternative? A prospective randomized study]. Unfallchirurg. 2000 Oct;103(10):826-33. doi: 10.1007/s001130050628. German. PMID 11098741
- [Background] Ludvigsen TC, Johansen S, Svenningsen S, Saetermo R. External fixation versus percutaneous pinning for unstable Colles' fracture. Equal outcome in a randomized study of 60 patients. Acta Orthop Scand. 1997 Jun;68(3):255-8. doi: 10.3109/17453679708996696. PMID 9246988
- [Background] Christensen OM, Kunov A, Hansen FF, Christiansen TC, Krasheninnikoff M. Occupational therapy and Colles' fractures. Int Orthop. 2001;25(1):43-5. doi: 10.1007/s002640000183. PMID 11374267
- [Background] Abbaszadegan H, Jonsson U, von Sivers K. Prediction of instability of Colles' fractures. Acta Orthop Scand. 1989 Dec;60(6):646-50. doi: 10.3109/17453678909149595. PMID 2624083
- [Background] MacDermid JC. Development of a scale for patient rating of wrist pain and disability. J Hand Ther. 1996 Apr-Jun;9(2):178-83. doi: 10.1016/s0894-1130(96)80076-7. No abstract available. PMID 8784681
- [Background] MacDermid JC, Turgeon T, Richards RS, Beadle M, Roth JH. Patient rating of wrist pain and disability: a reliable and valid measurement tool. J Orthop Trauma. 1998 Nov-Dec;12(8):577-86. doi: 10.1097/00005131-199811000-00009. PMID 9840793
- [Background] Stucki G, Liang MH, Phillips C, Katz JN. The Short Form-36 is preferable to the SIP as a generic health status measure in patients undergoing elective total hip arthroplasty. Arthritis Care Res. 1995 Sep;8(3):174-81. doi: 10.1002/art.1790080310. PMID 7654802
- [Background] MacDermid JC, Richards RS, Donner A, Bellamy N, Roth JH. Responsiveness of the short form-36, disability of the arm, shoulder, and hand questionnaire, patient-rated wrist evaluation, and physical impairment measurements in evaluating recovery after a distal radius fracture. J Hand Surg Am. 2000 Mar;25(2):330-40. doi: 10.1053/jhsu.2000.jhsu25a0330. PMID 10722826
- [Background] Jebsen RH, Taylor N, Trieschmann RB, Trotter MJ, Howard LA. An objective and standardized test of hand function. Arch Phys Med Rehabil. 1969 Jun;50(6):311-9. No abstract available. PMID 5788487
- [Background] MacDermid JC, Donner A, Richards RS, Roth JH. Patient versus injury factors as predictors of pain and disability six months after a distal radius fracture. J Clin Epidemiol. 2002 Sep;55(9):849-54. doi: 10.1016/s0895-4356(02)00445-6. PMID 12393071
- [Background] Swiontkowski MF, Engelberg R, Martin DP, Agel J. Short musculoskeletal function assessment questionnaire: validity, reliability, and responsiveness. J Bone Joint Surg Am. 1999 Sep;81(9):1245-60. doi: 10.2106/00004623-199909000-00006. PMID 10505521
- [Background] Friberg S, Lundstrom B. Radiographic measurements of the radio-carpal joint in normal adults. Acta Radiol Diagn (Stockh). 1976 Mar;17(2):249-56. doi: 10.1177/028418517601700212. PMID 1274658
- [Background] Taleisnik J, Watson HK. Midcarpal instability caused by malunited fractures of the distal radius. J Hand Surg Am. 1984 May;9(3):350-7. doi: 10.1016/s0363-5023(84)80222-1. PMID 6725893